CLINICAL TRIAL: NCT04334512
Title: A Randomized, Double-Blind, Placebo-Controlled Phase IIa Study of Quintuple Therapy to Treat COVID-19 Infection
Brief Title: A Study of Quintuple Therapy to Treat COVID-19 Infection
Acronym: HAZDpaC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ProgenaBiome (Other)
Collaborators: DSCS CRO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRG-044
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: COVID-19; Corona Virus Infection; Coronavirus-19; Sars-CoV2
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Hydroxychloroquine; Azithromycin; Ascorbic Acid; Vitamin D; Zinc

STUDY DESIGN:
Intervention Model Description: This is a Randomized, Double-Blind, Placebo-Controlled Phase II interventional Study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quintuple Therapy (Experimental): Patients will be treated with quintuple therapy for 10 days.
  Interventions: Drug: Hydroxychloroquine; Drug: Azithromycin; Dietary Supplement: Vitamin C; Dietary Supplement: Vitamin D; Dietary Supplement: Zinc
- Placebo (Placebo Comparator): Patients will be treated with placebo.
  Interventions: Dietary Supplement: Vitamin C; Dietary Supplement: Vitamin D; Dietary Supplement: Zinc

INTERVENTIONS:
Drug: Hydroxychloroquine — Treatment with hydroxychloroquine
  Other Names: Plaquenil
  Arms: Quintuple Therapy
Drug: Azithromycin — Treatment with azithromycin
  Other Names: Zithromax
  Arms: Quintuple Therapy
Dietary Supplement: Vitamin C — Treatment with vitamin C
Dietary Supplement: Vitamin D — Treatment with vitamin D
Dietary Supplement: Zinc — Treatment with Zinc

SUMMARY:
This is a Phase II interventional study will test the efficacy of quintuple therapy (Hydroxychloroquine, Azithromycin, Vitamin C, Vitamin D, and Zinc) in the treatment of patients with COVID-19 infection).

DETAILED DESCRIPTION:
In this study patients will be treated with a combination therapy to determine if this combination can effectively treat COVID-19. Treatment will last ten days. The study will last 24 weeks.

ELIGIBILITY:
1. Informed consent provided electronically via the EDC, demonstrating that the subject understands the procedures required for the study and the purpose of the study
2. Male or female subjects 18 years of age and up
3. Subjects must agree to practice at least two highly effective methods of birth control for the duration of the study. This includes condoms with spermicide, oral birth control pills, contraceptive implants, intra-uterine devices, or diaphragms. At least one of these must be a barrier method. Subjects not of reproductive potential will be exempt (e.g. post-menopausal, surgically sterilized)
4. Diagnosis of COVID-19 by RT-PCR

Exclusion Criteria

1. Refusal to provide informed consent
2. Diarrhea prior to infection
3. Any comorbidities which, in the opinion of the investigator, constitute health risk for the subject
4. Any contraindications for treatment with hydroxychloroquine

   1. Hypoglycemia
   2. Known G6PD deficiency
   3. Porphyria
   4. Anemia
   5. Neutropenia
   6. Alcoholism
   7. Myasthenia gravis
   8. Skeletal muscle disorders
   9. Maculopathy
   10. Changes in visual field
   11. Liver disease
   12. Psoriasis
5. Anemia from pyruvate kinase and G6PD deficiencies
6. Abnormal EKG with QT prolongation acquired or from birth
7. Allergies to 4-Aminoquinolines
8. History of jaundice or high fevers prior to developing COVID-19
9. Treatment with any of the medications listed in Appendix II
10. Treatment with any other drug not listed that affects the QT interval
11. Treatment with any anti-epileptic drug, whether prescribed for seizures or otherwise.
12. Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
The rate of recovery of mild or moderate COVID-19 in patients using Quintuple Therapy | 12 weeks
  Number of days from COVID-19 diagnosis to recovery via RT-PCR
Reduction or Progression of Symptomatic Days | 12 weeks
  Reduction and/or progression of symptomatic days, reduction of symptom severity
Assess the safety of Quintuple Therapy | 12 weeks
  Assess the symptom response to study therapy as measured by the survey in the EDC
Assess the safety of Quintuple Therapy via pulse | 12 weeks
  Pulse from baseline to 12 weeks
Assess the safety of Quintuple Therapy via oxygen saturation | 12 weeks
  Oxygen saturation from baseline to 12 weeks
Assess the safety of Quintuple Therapy via EKG | 12 weeks
  EKG response from baseline to 12 weeks
Assess Tolerability of Quintuple Therapy | 12 weeks
  Assess Adverse Events and Serious Adverse Events due to Quintuple Therapy

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Hazan, MD, Principal Investigator — ProgenaBiome
Locations (1):
- ProgenaBiome, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banjanac M, Munic Kos V, Nujic K, Vrancic M, Belamaric D, Crnkovic S, Hlevnjak M, Erakovic Haber V. Anti-inflammatory mechanism of action of azithromycin in LPS-stimulated J774A.1 cells. Pharmacol Res. 2012 Oct;66(4):357-62. doi: 10.1016/j.phrs.2012.06.011. Epub 2012 Jul 3. PMID 22766077
- [Background] Cortegiani A, Ingoglia G, Ippolito M, Giarratano A, Einav S. A systematic review on the efficacy and safety of chloroquine for the treatment of COVID-19. J Crit Care. 2020 Jun;57:279-283. doi: 10.1016/j.jcrc.2020.03.005. Epub 2020 Mar 10. PMID 32173110
- [Background] Gao J, Tian Z, Yang X. Breakthrough: Chloroquine phosphate has shown apparent efficacy in treatment of COVID-19 associated pneumonia in clinical studies. Biosci Trends. 2020 Mar 16;14(1):72-73. doi: 10.5582/bst.2020.01047. Epub 2020 Feb 19. PMID 32074550
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Background] Zhang L, Liu Y. Potential interventions for novel coronavirus in China: A systematic review. J Med Virol. 2020 May;92(5):479-490. doi: 10.1002/jmv.25707. Epub 2020 Mar 3. PMID 32052466